CLINICAL TRIAL: NCT00572754
Title: Phase II Trial to Evaluate the Safety and Efficacy of the Dry Circumcision
Brief Title: Phase II Trial to Evaluate the Safety and Efficacy of the Dry Circumcision Method
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Progressus (Other)
Responsible Party: Bertran Auvert, University of Versailles (France)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Drycirc Vz10d; NEB002180
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Circumcision; Male
MeSH Terms: interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Circumcision — Circumcision by tying a ligature around the foreskin.

SUMMARY:
The objective of this clinical investigation is to provide the first and preliminary clinical data to study the safety and efficacy of male circumcision where the dry circumcision method is employed.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects, aged 21 years or above at the point of screening for participation.
2. Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
3. Subjects who, in the opinion of the clinical investigator, are able to understand this clinical investigation co-operate with the investigational procedures and are willing to return to the clinical centre for all the required post-treatment follow-ups.
4. Subjects willing to be circumcised for cultural reasons.
5. Subjects living in the site's area.
6. Subjects who can be easily contacted by telephone.
7. Subjects who can correctly speak and correctly read English.

Exclusion Criteria:

1. Subjects who, in the opinion of the investigator, have an existing condition that would compromise their participation and follow-up in this study.
2. Subjects who are circumcised (i.e. subjects with a foreskin unable to cover the entire glans without pulling on the foreskin).
3. Subjects with a disease which is an indication for circumcision: phimosis, paraphimosis, warts under the prepuce, torn or tight frenulum.
4. Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.
5. Subjects who have participated in a clinical study with an investigational product in the last 6 months.
6. Subjects who have an abnormal penile anatomy.
7. Subjects who are currently involved in any injury litigation claims.
8. Subjects who have penile diseases or lesions.
9. Subjects who have clinical symptoms of sexually transmitted infections.
10. Subjects with opportunistic infections.
11. Subjects with known diabetes, known allergy to local anaesthesia or with known abnormal blood coagulation.
12. Subjects whose penile circumference is higher (>3mm) or lower (<3mm) than the available circumcision tubes.
13. Subjects with a thick foreskin (difference between the diameter of covered glans and uncovered glans > 5mm).

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-11; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
The operative and short-term post-operative safety rates | 1 month

SECONDARY OUTCOMES:
Mobibidity and mortality The length of the residual foreskin. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Bertran Auvert, MD, PhD, Principal Investigator — UVSQ-INSERM-France
Locations (1):
- University Teaching Hospital, Lusaka, Zambia